CLINICAL TRIAL: NCT00241878
Title: Preschool Based Obesity Prevention Effectiveness Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Eric Gislason, Office of Research Services, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 334; R01HL081645 (NIH)
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2007-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

ARMS (2):
- 1 (Experimental): Teacher-Delivered Weight Control Intervention
  Interventions: Behavioral: Teacher-Delivered Weight Control Intervention
- 2 (Other): Teacher-Delivered General Health Intervention
  Interventions: Behavioral: Teacher-Delivered General Health Intervention

INTERVENTIONS:
Behavioral: Teacher-Delivered Weight Control Intervention — The teacher-delivered weight control intervention (TD-WCI) is implemented over 14 weeks with three lessons per week. Many lessons include the use of colorful, friendly, hand-made puppets that represent the seven food groups of the food pyramid (Miss Grain, Miss Fruit, Mr. Vegetable, Mr. Protein, Miss Dairy, Mr. Fat and Miss Sugar). Please see Appendix IX for complete curriculum and pictures of puppets. There are three 40-minute lessons per week that consist of a 15-20 minutes interactive healthy eating and exercise didactic session and then 20 minutes of ongoing physical activity (5 minutes warm-up, 15 minutes aerobic activity composed of a number of games and dances with music, 5 minutes cool-down). In addition to the child-based curriculum the WCI has parent newsletters. These newsletters are distributed on a weekly basis and provide information that parallels the children's curriculum
  Arms: 1
Behavioral: Teacher-Delivered General Health Intervention — The teacher-delivered general health intervention (TD-GHI) serves as the control group in the proposed study. TD-GHI is a general health intervention that is similar in structure and length to TD-WCI. Topics include those related to general health and safety, such as car safety, being a good friend, poison safety, disease prevention, etc. An example of an activity is the 911 emergency call. The children learn what 911 is and what would be an appropriate call. They then practice calling 911 on play telephones and relating the important information: nature of the emergency, their name, their address, etc. They learn also to stay on the phone with the 911 dispatcher until someone comes to help them. In addition to the child-based curriculum the GHI has parent newsletters. Like TD-WCI these newsletters are distributed on a weekly basis and provide information that parallels the children's curriculum
  Arms: 2

SUMMARY:
The purpose of this study is to compare changes in body mass index (BMI) among 3- to 5-year-old minority children randomized to a weight control intervention (WCI) or a general health control intervention.

DETAILED DESCRIPTION:
BACKGROUND:

Obesity is epidemic in the U.S. and is associated with increased risk for numerous medical problems. Many obesity-related risk factors are strikingly apparent in minority populations. Ethnic differences in obesity related risk factors begin as early as six to nine years of age. Thus, the need for overweight prevention efforts as early as the preschool years is critical.

This study builds upon the findings of the "Hip-Hop to Health" program. The primary aim of Hip-Hop was to compare changes in body mass index (BMI [kg/m2]) in two groups of 3- to 5-year-old minority children randomized to a Weight Control Intervention (WCI) or a General Health Control Intervention (GHI). Results for the children at the Year 1 and 2 follow-ups showed that children in the WCI had significantly smaller relative changes in BMI compared to children in the GHI control group. The success was among the schools that served predominantly Black children. Hip-Hop to Health was an efficacy trial delivered by trained specialists in early childhood education, and the first efficacy trial to document change in BMI in preschool children.

DESIGN NARRATIVE:

This study will test a 14-week teacher-delivered weight control intervention (TD-WCI) to a 14-week teacher delivered general health control intervention (TD-GHI) in a randomized community trial occurring in 16 preschools in the Chicago School District. The study has the following aims: 1) to compare children in these two conditions on changes in BMI post intervention and at Year 1 follow-up; 2) to compare children in these two conditions on changes in television viewing, physical activity, and fat, fiber, fruit and vegetable intake at post-intervention and Year 1 follow-up; and 3) to compare classroom teachers in these two conditions on nutrition and exercise knowledge, nutrition attitudes, and support for healthy eating post-intervention and Year 1 follow-up.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Inclusion Criteria:

* Have received an annual physical
* Parent or guardian willing to give informed consent
* Parent or guardian willing to provide demographic and anthropometric data and agree to complete food intake and physical activity information for their child

Exclusion Criteria:

* Requires a specialized diet outside of that served by the Chicago Public Schools
* Has a chronic physical or behavioral disorder that requires participant to be under close medical psychological supervision and routinely absent from the study

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 648 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Body height and weight | Sept 2006- May 2009
Healthy Start Knowledge Quiz | Sept 2006- May 2009
24-hour diet observation and recall | Sept 2006- May 2009
Physical activity | Sept 2006- May 2009
Television viewing (child outcomes, measured immediately after the study and at a 1-year follow-up visit) | Sept 2006- May 2009
Score on short Acculturation Scale (parent outcome, measured immediately after the study and at a 1-year follow-up visit) | Sept 2006- May 2009
Nutrition and exercise knowledge | Sept 2006- May 2009
Self-efficacy for eating and exercise behaviors | Sept 2006- May 2009
Score on Nutrition Attitudes Scale | Sept 2006- May 2009
Support and role modeling for healthy eating (teacher outcomes, measured immediately after the study and at a 1-year follow-up visit) | Sept 2006- May 2009

CONTACTS AND LOCATIONS:
Overall Officials: Marian Fitzgibbon, Principal Investigator — University of Illinois at Chicago

REFERENCES:
- [Derived] Kong A, Buscemi J, Stolley MR, Schiffer LA, Kim Y, Braunschweig CL, Gomez-Perez SL, Blumstein LB, Van Horn L, Dyer AR, Fitzgibbon ML. Hip-Hop to Health Jr. Randomized Effectiveness Trial: 1-Year Follow-up Results. Am J Prev Med. 2016 Feb;50(2):136-44. doi: 10.1016/j.amepre.2015.07.008. Epub 2015 Sep 16. PMID 26385162